CLINICAL TRIAL: NCT00070096
Title: A Phase II Study of BMS-247550 In Advanced Germ Cell Tumor Patients - THERAPEUTIC/DIAGNOSTIC PROTOCOL
Brief Title: Ixabepilone in Treating Patients With Advanced Cisplatin-Refractory Germ Cell Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000329992; MSKCC-03041; NCI-6022
Record Dates: First submitted 2003-10-03; First posted 2003-10-07 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2006-04

CONDITIONS: Brain and Central Nervous System Tumors; Extragonadal Germ Cell Tumor; Ovarian Cancer; Testicular Germ Cell Tumor
Keywords: stage IV ovarian germ cell tumor; recurrent ovarian germ cell tumor; adult central nervous system germ cell tumor; recurrent malignant testicular germ cell tumor; stage III malignant testicular germ cell tumor; testicular seminoma; testicular choriocarcinoma and embryonal carcinoma; testicular choriocarcinoma and seminoma; testicular choriocarcinoma and teratoma; testicular choriocarcinoma and yolk sac tumor; testicular choriocarcinoma; testicular embryonal carcinoma and seminoma; testicular embryonal carcinoma and teratoma with seminoma; testicular embryonal carcinoma and teratoma; testicular embryonal carcinoma and yolk sac tumor with seminoma; testicular embryonal carcinoma and yolk sac tumor; testicular embryonal carcinoma; testicular yolk sac tumor and teratoma with seminoma; testicular yolk sac tumor and teratoma; testicular yolk sac tumor; recurrent extragonadal non-seminomatous germ cell tumor; recurrent extragonadal seminoma; stage IV extragonadal non-seminomatous germ cell tumor; stage IV extragonadal seminoma; recurrent extragonadal germ cell tumor; testicular immature teratoma; testicular mature teratoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Ovarian Neoplasms; Testicular Germ Cell Tumor; Testicular Neoplasms; Seminoma; Carcinoma, Embryonal; Teratoma; Endodermal Sinus Tumor | interventions — ixabepilone

INTERVENTIONS:
Drug: ixabepilone

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as ixabepilone, work in different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: This phase II trial is studying how well ixabepilone works in treating patients with metastatic germ cell tumors that are refractory to cisplatin.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of ixabepilone in patients with metastatic cisplatin-refractory germ cell tumors.
* Determine the safety of this drug in these patients.

OUTLINE: Patients receive ixabepilone IV over 3 hours on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 10-29 patients will be accrued for this study within 1.3-4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed germ cell tumor (GCT) (seminoma or non-seminoma) meeting the following criteria:

  * Measurable metastatic disease by one of the following methods:

    * Radiography

      * If eligibility is defined by measurable disease only, there must be at least 1 site that has not been previously irradiated
    * Alpha-fetoprotein greater than 15 ng/mL and/or ß-human chorionic gonadotropin greater than 2.2 mIU/L
* Previously treated progressive disease meeting 1 of the following criteria:

  * Not a candidate for potentially curative therapy OR has already received high-dose chemotherapy regimens (prior paclitaxel allowed)
  * Deemed to be cisplatin-refractory after prior cisplatin-based regimen AND does not want to have potentially curative high-dose therapy (mediastinal or primary refractory GCT)
  * Prior treatment with 1 cisplatin-based regimen (primary mediastinal nonseminomatous GCT)

PATIENT CHARACTERISTICS:

Age

* 16 and over

Performance status

* Karnofsky 70-100%

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count greater than 100,000/mm^3
* Hemoglobin at least 10 g/dL

Hepatic

* Bilirubin no greater than 1.5 times normal
* SGOT no greater than 2 times upper limit of normal

Renal

* Creatinine no greater than 2.2 mg/dL

Other

* Not pregnant or nursing
* Negative pregnancy test
* No active infection

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent immunotherapy

Chemotherapy

* See Disease Characteristics
* No other concurrent cytotoxic chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* No concurrent radiotherapy

Surgery

* Not specified

Other

* No other concurrent experimental or commercial anticancer medications or therapies

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2003-08; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Efficacy
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Gnanamba V. Kondagunta, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States